CLINICAL TRIAL: NCT02828098
Title: An Exploratory First in Human Phase I Clinical and Pharmacokinetic Study of Intra-tumoral Administration of BO-112 in Adult Patients With Aggressive Solid Tumors, With an Extension Cohort in Combination With Anti-PD1 Treatment
Brief Title: Exploratory Study of BO-112 in Adult Patients With Aggressive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Highlight Therapeutics (Industry)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 112/2016-IT
Record Dates: First submitted 2016-06-23; First posted 2016-07-11 (Estimated); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: aggressive solid tumors
MeSH Terms: conditions — Neoplasms | interventions — spartalizumab

ARMS (2):
- Part 1: BO-112 IT (Experimental): BO-112 dose 1 (starting dose) intratumoral injection. BO-112 dose 2, 3 and 4 are expected to be tested, upon confirmation of the safety profile of the starting dose.
  Interventions: Drug: Part 1: BO-112
- Part 2: BO-112 IT (Experimental): Combination treatment of BO-112 intratumoral injections with standard of care nivolumab intravenous treatment
  Or Combination treatment of BO-112 intratumoral injections with standard of care pembrolizumab intravenous treatment
  Interventions: Drug: Part 2: BO-112

INTERVENTIONS:
Drug: Part 1: BO-112 — Cohorts of three patients per dose level will be treated consecutively in the absence of Dose Limiting Toxicity (DLT).
  Arms: Part 1: BO-112 IT
Drug: Part 2: BO-112 — BO-112 at a fixed dose will be administered as an intratumoral injection for up to 5 doses over 12 weeks and continue as long as there is benefit.
  Nivolumab will be administered as an intravenous infusion every 2 weeks at a dose of 3 mg/kg for up to a total period of one year.
  OR Pembrolizumab will be administered as an intravenous infusion every 3 weeks at either 200 mg or at 2 mg/kg depending on the indication, for up to a total period of one year.
  Other Names: anti-PD1 monoclonal antibody
  Arms: Part 2: BO-112 IT

SUMMARY:
Part 1: 16 to 32 patients with aggressive solid tumors from whom biopsies can be obtained, will receive BO-112 through IT administration.

Injected lesions must be palpable and biopsiable at the time of injection, and biopsied after 7-14 days. Patients will not receive an alternative therapy during the period comprising from first and second biopsy. BO-112 will be administered at a starting dose. Upon confirmation of the safety profile of the starting dose and evaluation of the pharmacokinetic (PK) profile, three additional dose levels are expected to be tested.

During the course of the study, subjects will be examined for any side effects that may occur (safety and tolerability).

Additionally this study will also study BO-112 biological activity, the innate and adaptive immune system response and signaling pathways, as well as signs of clinical relevance, will be studied.

Part 2: An additional 30 patients with progressive disease while on anti-PD1 treatment for an approved indication, will receive BO-112 through IT administration in combination with the anti-PD1 treatment to evaluate the safety and tolerability of the combination.

Injected lesions must be palpable and biopsiable at the time of injection. Patients will continue with their anti-PD1 treatment. During the course of the study, patients will be examined for any side effects that may occur (safety and tolerability).

Additionally this part of the trial will also study BO-112 biological activity, the innate and adaptive immune system response and signaling pathways, as well as signs of clinical response

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 years or more on the day of signing informed consent form.
2. Histologically or cytologically confirmed aggressive solid tumors
3. Patients must have:

   * Biopsy-accessible tumors
   * No prior anticancer treatment during the last 14 days

Additional inclusion criteria for Part 2: disease progression on treatment with anti-PD1 antibody for an approved indication

Exclusion Criteria:

Other relevant and clinically significant concomitant diseases or adverse clinical conditions which may jeopardize patient safety:

* Increased cardiac risk: congestive heart failure; or unstable angina pectoris; or arrhythmia requiring treatment or uncontrolled arterial hypertension; or myocardial infarction within 12 months before inclusion in the study.
* Patients with active central nervous system (CNS) lesions (including carcinomatous meningitis) will be excluded. However, patients will be eligible if:

  * All known CNS lesions have been treated with stereotactic therapy or surgery, AND
  * There has been no evidence of clinical and radiographic disease progression in the CNS for ≥ 4 weeks after radiotherapy or surgery, and has not required to increase in the last 4 weeks their steroids use or has not started a new course of steroids
  * Whole brain radiotherapy is not allowed, with the exception of patients who have had definitive resection or stereotactic therapy of all radiologically detectable parenchymal brain lesions.
* Active infection.
* Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis B or C).
* Any clinically significant abnormality on history or examination including diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication (physiologic doses of corticosteroids may be approved after consultation with the Sponsor).

Additional exclusion criteria for Part 2: Grade 3-4 toxicity due to anti-PD1 antibody or permanent discontinuation of anti-PD1 antibody due to immune related or other adverse reaction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-06; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Part 1: Day 30 after administration of the last dose. Part 2: 12 weeks and for patients who continue up to 1 year
  To evaluate the safety and tolerability of B0-112 in terms of adverse events at every visit

SECONDARY OUTCOMES:
Circulating cytokines including type I IFNs, TNFalpha and IL6 (by ELISA) | Part 1: At three independent points during the study. Day 7-1 prior to administration, 24 hours after administration and 7-14 days after administration of the agent. Part 2: 12 weeks
Plasma levels of BO-112 | Part 1: 0-15-30-240 minutes and 24 hours after administration of the drug. Part 2: 1 day
  To characterize the pharmacokinetics (PK) of BO-112 by measuring the amount in plasma at regular timepoints during the study
Anti-tumor activity | 12 weeks and for patients who continue up to 1 year
  Part 2 only: To evaluate the antitumor activity of the combination of BO-112 and anti-PD1 treatment

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Clínica Universitaria Navarra, Pamplona, Navarre
  - ICO Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Quiron Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga

REFERENCES:
- [Derived] Aznar MA, Planelles L, Perez-Olivares M, Molina C, Garasa S, Etxeberria I, Perez G, Rodriguez I, Bolanos E, Lopez-Casas P, Rodriguez-Ruiz ME, Perez-Gracia JL, Marquez-Rodas I, Teijeira A, Quintero M, Melero I. Immunotherapeutic effects of intratumoral nanoplexed poly I:C. J Immunother Cancer. 2019 May 2;7(1):116. doi: 10.1186/s40425-019-0568-2. PMID 31046839